CLINICAL TRIAL: NCT03890757
Title: Efficacy of Serratus Anterior Plane Block Versus Thoracic Paravertebral Block in Patients With Unilateral Multiple Rib Fractures: Comparative Randomized Study
Brief Title: Serratus Anterior Plane Block , Paravertebral Block and Quality of Analgesia in Patients With Blunt Chest Trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samaa Rashwan (Other)
Responsible Party: Sponsor-Investigator, Samaa Rashwan, Samaa Abou Alkassem Rashwan, Beni-Suef University
Organization: Beni-Suef University (Other)
Other Study IDs: Beni-Suef University Hospital
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- serratus anteriorblock: Serratus plane block will be performed with the patient in the lateral position and the arm abducted. Using a high-frequency linear ultrasound probe
  Interventions: Other: ultrasound guided paravertebral or serratus anterior block

INTERVENTIONS:
Other: ultrasound guided paravertebral or serratus anterior block — Patients groups will be as follow:
  Group (I): Serratus plane block will be performed with the patient in the lateral position and the arm abducted. Using a high-frequency linear ultrasound probe ,Group (II): thoracic paravertebral block will be performed in the sitting position. The spinal level chosen for needle insertion will be two segments below the upper most fractured rib or midway between the upper most and lowest fractured rib, 2-2.5 cm distance from the midline in the same injury site

SUMMARY:
Pain associated with rib movement cause inability to cough and breathe deeply that leads to reduction in the tidal volume and predisposes to significant atelectasis, sputum retention, pneumonia and a reduction in functional residual capacity .These factors in turn lead to decreased lung compliance, ventilation perfusion mismatch, hypoxemia and respiratory distress. Therefore, effective pain relief remains the cornerstone of management to prevent serious respiratory complications .

DETAILED DESCRIPTION:
Thoracic paravertebral block and other regional techniques like intrapleural block and intercostal nerve blocks have variable success and high potential for local anaesthetic toxicity. Serratus anterior plane block is relatively novel technique that is less invasive, easier to perform and improve pulmonary function that reduces the incidence of pneumonia, number of ventilator days, and mortality, especially those sustaining five or more rib fractures

ELIGIBILITY:
Inclusion Criteria:Patients aging from 20 to 70 years old.

* ASA physical status status I-II -- Patients suffering from blunt chest trauma with unilateral multiple rib fractures.

Exclusion Criteria:• Spinal cord injury.

* Epidural or spinal cord haematoma.
* Thoracic vertebral body fracture.
* Spinal injury awaiting assessment.
* Coagulopathy (platelets <50×109 litre-1, INR>1.5).
* Local infection or sepsis.
* Allergy to local anaesthetic.
* Inability to position patient due to associated injuries.
* Severe traumatic brain injury.
* Unstable lumbar or cervical spinal fractures.
* Hypotension.
* Hypovolaemia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult malesandfemales
Study Population: Patients aging from 20 to 70 years old. - ASA physical status status I-II
  -- Patients suffering from blunt chest trauma with unilateral multiple rib fractures.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study was to compare ultrasound guided serratus anterior plane block and ultrasound guided paravertebral block as regard the efficacy of analgesia in patients with blunt chest trauma with unilateral multiple rib fractures | VAS will be recorded before performing the technique , this will be the base line record, then it will be compared by the value of VAS 30 minutes after performing the technique and the value of VAS at 1, 3, 6,12 and 24 hours
  pain will be assessed by the visual analogue scale(VAS)

SECONDARY OUTCOMES:
total dose of rescue analgesia | the observation will be for 24 hours
  Analgesic requirement in the form of 25 mg pethidin intravenously if VAS score >3

CONTACTS AND LOCATIONS:
Overall Officials: Samaa Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No